CLINICAL TRIAL: NCT00135135
Title: Neuroblastoma Protocol 2005: Therapy for Children With Advanced Stage High-Risk Neuroblastoma
Brief Title: Therapy for Children With Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: AstraZeneca (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Wayne L. Furman M.D./Prinicipal Investigator, St.Jude Children's Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NB2005; AstraZeneca IRUSIERS0389
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-06

CONDITIONS: Neuroblastoma
Keywords: Cancer; Childhood Tumor; Neoplasms
MeSH Terms: conditions — Neuroblastoma; Neoplasms | interventions — Gefitinib; Irinotecan; Doxorubicin; Etoposide; Cisplatin; Topotecan; Carboplatin; Melphalan; Isotretinoin; Radiotherapy; Surgical Procedures, Operative; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Drug: Gefitinib, Irinotecan, Cycophosphamide, Doxorubicin, Etoposide, Cisplatin, Topotecan, Carboplatin, Melphalan, 13-cis retinoic acid; Procedure: Radiation therapy, Surgery, Peripheral Stem cell transplant

INTERVENTIONS:
Drug: Gefitinib, Irinotecan, Cycophosphamide, Doxorubicin, Etoposide, Cisplatin, Topotecan, Carboplatin, Melphalan, 13-cis retinoic acid — See Detailed Description.
Procedure: Radiation therapy, Surgery, Peripheral Stem cell transplant — See Detailed Description.

SUMMARY:
This is a phase II window study of the combination of ZD1839 (gefitinib) and irinotecan in children with high-risk neuroblastoma followed by standard induction chemotherapy, intensification with autologous stem cell transplantation, and an oral maintenance phase with 13-cis-retinoic acid and topotecan. We hypothesize that the ZD1839 (gefitinib) and irinotecan window will be efficacious.

DETAILED DESCRIPTION:
The study will have five parts or phases. In the first part the combination of irinotecan and gefitinib will be studied. After that, patients who have responded well will have surgery to remove the tumor. This will be followed by a third part which includes about nine months of treatment with cisplatin, adriamycin, etoposide, cyclophosphamide, and topotecan. The fourth part will be intensification with melphalan, etoposide and carboplatin and blood stem cell rescue. During this part, radiation will also be given to the sites of the disease. Finally, monthly treatments with oral retinoic acid, alternating with oral topotecan, will be continued for a total of 16 months of maintenance. It is anticipated that it will take about 2 years to complete this entire treatment plan.

This study has multiple therapeutic, pharmacologic, biologic, and diagnostic imaging objectives:

* To estimate whether oral gefitinib with two courses of intravenous irinotecan will decrease the incidence of fever/neutropenia, duration of hospitalization, duration of intravenous antibiotics and numbers of platelet and RBC transfusions during the first six weeks of treatment compared to the topotecan window in NB97.
* To estimate local control of primary site disease to this treatment plan.
* To estimate the overall survival and progression-free survival in patients treated with this approach.
* To estimate the feasibility of resecting the primary tumor after two courses of irinotecan and gefitinib.
* To evaluate the disposition of irinotecan and gefitinib in previously untreated patients with neuroblastoma.
* To evaluate the disposition of intravenous and oral topotecan in previously untreated patients with neuroblastoma.
* To evaluate the pharmacogenetic determinants of gefitinib and irinotecan pharmacokinetics and pharmacodynamics (e.g., CYP3A4/5, UGT1A1, and ABCG2 (BCRP) polymorphisms).
* To evaluate the pharmacogenetic determinants of topotecan pharmacokinetics and pharmacodynamics (e.g., CYP3A4/5 and ABC transporter polymorphisms).
* To evaluate in tumor samples the molecular and cellular expression of EGFR, MRP4 and ABCG2 (BCRP) utilizing appropriate laboratory techniques.
* To describe the relative frequency of positive bone marrow by sensitive MRD methods at diagnosis, after window therapy, at the time of stem cell harvest, and at several time points following the completion of intensification. These results will be compared with timing and pattern of disease recurrence.
* To describe what percentage of primary or metastatic neuroblastomas have amplified ICAM-2 and chromosome 17.
* To generate preliminary data regarding the potential use of ICAM-2 copy number as a prognostic indicator in neuroblastoma.
* To determine the levels of the angiogenic factors VEGF and bFGF in the peripheral circulation of patients at diagnosis, after window therapy, at the time of stem cell harvest and at several time points following the completion of intensification. These results will be compared with the degree of tumor response and the timing of disease recurrence.
* To procure tumor samples for construction of tissue microarray blocks that will be utilized in further biologic characterization of these tumors.
* To prospectively evaluate FDG PET imaging as a marker of disease at diagnosis, (pre and post window therapy), prior to intensification, and at the completion of therapy.
* To generate preliminary data on the use of contrast enhanced ultrasound and magnetic resonance imaging to evaluate changes in tumor vascularity at various timepoints in therapy.

Details of Treatment Interventions:

Window Phase Irinotecan 15mg/m2 daily x 5 days for two weeks with daily oral gefitinib 112.5 mg/m2 daily x 12 days., followed by 9 day rest, then same course repeated. Subjects that respond to window therapy receive the same course again instead of topotecan for Block 2, course 6 (week 21) of induction.

Induction Therapy (following window):

Cyclophosphamide 1.5 gm/m2 daily x 2 I.V. day 1 & 2 Adriamycin 50 mg/m2 I.V. day 1 only MESNA: 375 mg/m2 I.V. immediately following cyclophosphamide and at 3 and 6 hours post-infusion.

Etoposide: 30 mg/m2 over 30 minutes, followed by etoposide 250 mg/m2/day x 3 days I.V. by continuous infusion (days 2-5), given during induction therapy courses 1, 4, and 7.

Cisplatin 40 mg/m2/day x 5 I.V. over 1 hour (days 1-5) Etoposide 200 mg/m2/day x 3 I.V. over 1 hour (days 2, 3, 4), given during induction courses 2, 5, and 8.

IV topotecan adjusted to AUC 100 ± 20nghr/ml daily x 5 days for two weeks, during courses 3, 6 (for patients that do not respond to window), and 9 of induction.

Intensification:

Melphalan, Etopophos and carboplatin:Day -8, -7, -6, -5: Melphalan 45 mg/m2 IV Day -4: Etopophos 40 mg/kg/day IV Day -4, -3, & -2: Carboplatin (AUC target 4.1) Day 0- infusion of peripheral blood stem cells previously harvested by pheresis.

Maintenance:

13 cis-retinoic acid and oral topotecan courses:13-cis-retinoic acid 160 mg/m2/day divided into two equal doses given orally BID x 14 days, followed by a 14 day rest. This will be repeated x one. Subjects less or equal to 12 kg will be given 5.33 mg/kg/day divided BID. These courses are alternated with 2 months of oral topotecan once daily for 5 days for 2 consecutive weeks at 1.8 mg/m2/day , or 0.06 mg/kg/day for patients less than 12 months old (total of 10 doses) for a total of 16 courses (four, two-month courses of each).

Radiation therapy : Radiation therapy to the primary and metastatic disease sites will follow peripheral blood stem cell transplant with the exception of any patient requiring emergent radiation. External beam radiotherapy will be delivered to the primary site and select metastatic sites. Radiotherapy is planned to be initiated four weeks following stem cell reinfusion.

Surgery : After recovery from induction and re-evaluation of tumor status, subjects undergo surgery for resection of the primary tumor mass and careful lymph node staging, if surgery was not possible after the irinotecan and ZD1839 window.

Peripheral blood stem cell collection and infusion : After course 3, subjects undergo peripheral blood stem cell (PBSC) harvest. If this is unsuccessful, harvesting will be done with subsequent chemotherapy courses. Subjects are mobilized with filgrastim (10mcg/kg/day). PBSC harvesting will be performed by leukapheresis if possible, bone marrow harvest if not. Stem cells are stored and re-infused after intensification chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is less than or equal to 18 years of age
* Patient is newly diagnosed with high-risk neuroblastoma
* Patient has adequate kidney and liver function
* No prior therapy, unless an emergency situation requires local tumor treatment (discuss with PI)

Exclusion Criteria:

* Known severe hypersensitivity to ZD1839 or any of the excipients of this product
* Any evidence, as judged by the investigator, of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
* Evidence of any significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the trial.
* Pregnant or breast feeding (women of child-bearing potential).
* Concomitant use of phenytoin, carbamazepine, rifampicin, barbiturates, or St. John's Wort.
* Treatment with a non-approved or investigational drug within 30 days before Day 1 of study treatment.
* Any evidence of clinically active interstitial lung disease (patients with chronic stable radiographic changes who are asymptomatic need not be excluded).
* Children with INSS 4 disease, age <12 months with all 3 favorable biologic features (non-amplified MYCN, favorable pathology and DNA index

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2005-08; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Response rate | Within 30 days of completion of window therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne L Furman, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org